CLINICAL TRIAL: NCT06342297
Title: Dermatoscopy Guided Resection Margins in Basal Cell Carcinoma and Cutaneos Squamous Cell Carcinoma
Brief Title: Dermatoscopy Guided Resection for Skin Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Örebro County (Other)
Responsible Party: Principal Investigator, Fredrik Landström, Associate professor, Region Örebro County
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OLL-1003043
Record Dates: First submitted 2024-03-26; First posted 2024-04-02 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Basal Cell Carcinoma; Cutaneous Squamous Cell Carcinoma; Surgical Margin
Keywords: Dermatoscopy
MeSH Terms: conditions — Carcinoma, Basal Cell; Margins of Excision | interventions — Dermoscopy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No dermatoscopy (No Intervention): Dermatoscopy not used in decision of surgical margin
- Dermatoscopy (Experimental): Dermatoscopy is used in decision of surgical margin
  Interventions: Device: Dermatoscopy

INTERVENTIONS:
Device: Dermatoscopy — Dermatoscopy used in decision of surgical margin before resection of basal cell carcinoma or cutaneous squamous cell carcinoma
  Arms: Dermatoscopy

SUMMARY:
In this randomizid controlled trial the aim is to use dermatoscopy in deciding the resection margin for patients with suspected or verified basal cell carcinoma or cutaneous squamous cell carcinoma. The outcome is radical/non radical resection of the lateral margins in the pathology report.

DETAILED DESCRIPTION:
In basal cell carcinoma and especially cutaneous squamous cell carcinoma the prognosis is very good if the tumour is radically removed in the primary resection. In this study we propose that the use of dermatoscopy in deciding the surgical margins can increase the proportion of radically removed tumours. In this randomized clinical trial the use of dermatoscopy in deciding the surgical margins in patients with suspected or verified basal cell carcinoma or cutaneous squamous cell carcinoma is assessed. The outcome measure is radical/non radical resection of the lateral margins. In the control group dematoscopy is not used in deciding the surgical margin. 400 patients with suspected or verified BCC or cSCC will be included, 200 in each group.

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary suspected or verified basal cell carcinoma or cutaneous cell carcinoma

Exclusion Criteria:

* Recurrent tumours
* Previous radiotherapy of the tumour area
* If the patient cannot understand the study i nformation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-01-14 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2026-01-14 (Estimated)

PRIMARY OUTCOMES:
Pathology resection side margin (radical/not radical) | Pathology report usually within two weeks after surgery
  If the side margins in the pathology report is radical or not

CONTACTS AND LOCATIONS:
Locations (1):
- Örebro University Hospital, Örebro, Sweden